CLINICAL TRIAL: NCT01999686
Title: Polycystic Ovary Syndrome Treatment Using DLBS3233, Metformin, and Combination of Both, and Its Relation to Fertility
Brief Title: PCOS Treatment Using DLBS3233, Metformin, and Combination of Both
Acronym: POSITIF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS3233-1013
Record Dates: First submitted 2013-11-26; First posted 2013-12-03 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2019-05

CONDITIONS: Polycystic Ovary Syndrome (PCOS); Insulin Resistance
Keywords: Polycystic ovarium syndrome; DLBS3233; metformin; insulin resistance; Female
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance | interventions — DLBS3233

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment I : DLBS3233 (Experimental): DLBS3233 100 mg capsule once daily, and Placebo metformin caplet twice daily; orally, for 6 months
  Interventions: Drug: DLBS3233; Drug: Placebo metformin
- Treatment II : Metformin (Active Comparator): Metformin XR 750 mg caplet twice daily, and Placebo DLBS3233 once daily; orally, for 6 months
  Interventions: Drug: Metformin XR; Drug: Placebo DLBS3233
- Treatment III : Combination DLBS3233 and Metformin (Experimental): DLBS3233 100 mg capsule once daily, and Metformin XR 750 mg caplet twice daily; orally, for 6 months.
  Interventions: Drug: DLBS3233; Drug: Metformin XR

INTERVENTIONS:
Drug: DLBS3233
  Other Names: Inlacin
  Arms: Treatment I : DLBS3233; Treatment III : Combination DLBS3233 and Metformin
Drug: Metformin XR
  Other Names: Glumin XR
  Arms: Treatment II : Metformin; Treatment III : Combination DLBS3233 and Metformin
Drug: Placebo metformin — Placebo metformin has the same ingredients with Metformin XR caplet, except that it does not contain the active substance (metformin).
  Arms: Treatment I : DLBS3233
Drug: Placebo DLBS3233 — Placebo DLBS3233 has the same ingredients with DLBS3233 capsule, except that it does not contain the active substance (DLBS3233).
  Arms: Treatment II : Metformin

SUMMARY:
This is a 3-arm, randomized, double-blind, double-dummy, and controlled clinical study over 6 months of treatment to evaluate the metabolic and clinical efficacy as well as the safety of DLBS3233 alone, metformin and combination of both, in improving metabolic and reproductive parameters.

DETAILED DESCRIPTION:
There will be 3 groups of treatment (N = 186), each consist of 62 subjects, as the following:

* Treatment I : DLBS3233 100 mg once daily
* Treatment II : Metformin XR 750 mg twice daily
* Treatment III : DLBS3233 100 mg once daily and Metformin XR 750 mg twice daily.

Laboratory examination to evaluate metabolic efficacy parameters will be performed at baseline, Month 3rd, and end of study (Month 6th).

Clinical and laboratory examination to evaluate the reproductive efficacy parameters using trans-vaginal USG and biomarkers (such as reproductive hormones) will be performed at baseline to the end of study.

Safety examination will be performed at baseline and end of study. Occurrence of adverse event will be observed along the study conduct.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent prior to participation in the study.
2. Female subjects in reproductive age (i.e. 18-40 years) willing to conceive.
3. Subject with a diagnosis of polycystic ovary syndrome confirmed by two of the following (Rotterdam Criteria):

   * Hyperandrogenism (defined by elevated free testosterone concentration; or Ferriman-Gallwey Score of ≥ 8).
   * Ovarian dysfunction indicated by menstrual irregularity: oligomenorrhea (cycles of > 35 days), or amenorrhea (no menses in the last of 3 months) after negative screening pregnancy test.
   * Polycystic ovary as shown by ultrasonography (USG).
4. Subject with insulin resistance defined by : HOMA-IR of > 2.00.
5. Subject with body mass index (BMI) of 19-35 inclusive.
6. Able to take oral medication.

Exclusion Criteria:

1. Pregnant or lactating women (urinary pregnancy test will be applied at screening).
2. Based on previous or current medical (either laboratory or clinical) examination, subjects known to have any of the following conditions:

   * Cushing's syndrome, late onset of congenital adrenal hyperplasia, androgen-secreting tumors, uncontrolled thyroid disease, hyperprolactinemia.
3. Known to have the following medical condition:

   * Diabetes mellitus,
   * Uncontrolled hypertension
   * Symptomatic cardiovascular diseases:
   * Acute or chronic infections at baseline.
   * Any known malignancies.
4. History of gynecological surgery.
5. Impaired renal function
6. Impaired liver function
7. Medically-assisted weight loss with medications or surgical procedures.
8. Currently having laparoscopic ovarian diathermy (LOD).
9. Currently under treatment with in vitro fertilization (IVF) techniques.
10. Have been regularly taking any of the following medications, within ≤ 3 months prior to screening, such as:

    * Clomiphene citrate
    * Insulin sensitizers, i.e. metformin and thiazolidinediones
    * Aromatase inhibitors, such as: anastrozole, letrozole
    * Glucocorticoids
    * Gonadotropins
    * Gonadotropin-releasing hormone agonists (GnRHa)
    * Oral contraceptive pills (OCPs)
    * Antiandrogens, such as: spironolactone, cyproterone acetate (CPA), and flutamide
    * Any traditional or herbal medicines
11. Participating in other clinical trial within 30 days prior to screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2014-10; Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
HOMA-IR reduction | 6 months
  HOMA-IR reduction from baseline to Month 6th (end of study)

SECONDARY OUTCOMES:
Lipid profile improvement | 3 and 6 months
  Lipid profile improvement (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides level) from baseline to Month 3rd and Month 6th (end of study)
Improvement of glucose tolerance | 3 and 6 months
  Improvement of glucose tolerance (reduction of FPG and 2-hour PPPG) from baseline to Month 3rd and Month 6th (end of study)
Change of waist circumference | 1, 2, 3, 4, 5, and 6 months
  1, 2, 3, 4, 5, and 6 months
Response rate: presence of ovulation | menstrual cycle of Month 3rd up to that of Month 6th
  Presence of ovulation will be evaluated using trans-vaginal USG to find dominant follicle(s), at the day/period of ovulation, starting from menstrual cycle of Month 3rd up to Month 6th. Measurement of progesterone level will be performed 7 days after the finding of dominant follicle on USG examination to confirm the presence of ovulation.
Change of endometrium thickness | 3 to 6 months
  Change of endometrium thickness will be measured by using trans-vaginal USG at basal condition and at the day/period of ovulation
Improvement of S/A ratio | 3 to 6 months
  Improvement from baseline of the S/A ratio (defined as the ratio between stromal and total area of median ovarian section) will be measured using trans-vaginal USG (trans-longitudinal measurement) at Baseline, menstrual cycle of Month 3rd, and menstrual cycle of Month 6th at basal condition.
Improvement in Ferriman-Gallwey Score | 3 and 6 months
  Improvement in Ferriman-Gallwey Score from baseline to Month 3rd and Month 6th (the end of study)
Reduction of free testosterone level | 6 months
  Reduction of free testosterone level from baseline to Month 6th (end of study)
Change of luteinizing hormone (LH) level | 6 months
  Change of luteinizing hormone (LH) level from baseline to Month 6th (end of study)
Change of luteinizing hormone (LH) / follicle stimulating hormone (FSH) ratio | 6 months
  Change of luteinizing hormone (LH) / follicle stimulating hormone (FSH) ratio from baseline to Month 6th (end of study)
Liver function | 6 months
  Liver function (levels of serum AST, ALT, alkaline phosphatase) will be measured at baseline and Month 6th (end of study)
Renal function | 6 months
  Renal function (levels of serum creatinine, BUN) will be measured at baseline and Month 6th (end of study)
Number of adverse events and subjects with events | During 6 months
  Adverse events as well as number of events and subjects experiencing the events will be observed and evaluated throughout study period (6 months) and until all adverse events have been recovered or stabilized

CONTACTS AND LOCATIONS:
Overall Officials: Soehartono Ds, Prof. dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Airlangga, Dr. Soetomo Hospital, Surabaya, Indonesia.; Arsana Wiyasa IW, Dr. dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Brawijaya, Dr. Saiful Anwar Hospital, Malang, Indonesia.; Putu Doster Mahayasa, dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Udayana, Sanglah Hospital, Denpasar, Indonesia.; Syarief Taufik, dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, Diponegoro University, Dr. Kariadi Hospital, Semarang, Indonesia.; Nusratuddin Abdullah, Dr. dr., SpOG-K, MARS, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Hasanuddin, Dr. Wahidin Sudirohusodo Hospital, Makasar, Indonesia.; Iwan Darma Putra, dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Lambung Mangkurat, Ulin Banjarmasin Hospital, Banjarmasin, Indonesia.; Eddy Suparman, Prof. Dr. dr., SpOG-K, Principal Investigator — Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Sam Ratulangi, Prof. Dr. Kandou Hospital, Manado, Indonesia.
Locations (7):
- Indonesia (7):
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Lambung Mangkurat, Ulin Banjarmasin Hospital, Banjarmasin
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Udayana, Sanglah Hospital, Denpasar
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Hasanuddin, Dr. Wahidin Sudirohusodo Hospital, Makasar
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Brawijaya, Dr. Saiful Anwar Hospital, Malang
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Sam Ratulangi, Prof. Dr. Kandou Hospital, Manado
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, Diponegoro University, Dr. Kariadi Hospital, Semarang
  - Division of Reproductive Endocrinology and Infertility, Department of Obstetrics and Gynecology, Faculty of Medicine, University of Airlangga, Dr. Soetomo Hospital., Surabaya

REFERENCES:
- [Derived] Hidayat ST, Mulyantoro I, Damas S, Tjandrawinata RR. The Effect and Safety Assessment of Metformin and DLBS3233 (A Bioactive Fraction of Lagerstroemia speciosa and Cinnamomum burmannii) on Improving Metabolic Parameters in Women with Polycystic Ovary Syndrome. Int J Womens Health. 2023 Jul 4;15:971-985. doi: 10.2147/IJWH.S409685. eCollection 2023. PMID 37424700